CLINICAL TRIAL: NCT06396299
Title: COhort of antithrOmbotic Use and cLinical Outcomes in Patients With Atrial Fibrillation (COOL-AF) Phase 2
Status: Recruiting | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: Health Systems Research Institute,Thailand (Other Government); The Heart Association of Thailand (Unknown)
Responsible Party: Principal Investigator, Rungroj Krittayaphong, Professor, Mahidol University
Other Study IDs: COA-CREC103-2023
Record Dates: First submitted 2024-04-19; First posted 2024-05-02 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; ischemic stroke; major bleeding; death; oral anticoagulant
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke; Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients diagnosed with atrial fibrillation
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Atrial fibrillation (AF) is a leading cause of cardiovascular mortality and morbidity. Asian patients with AF have a higher rate of major bleeding including intracranial hemorrhage (ICH) compared to non-Asians. Non-vitamin K antagonist oral anticoagulants (NOACs) are the safer drugs compared to warfarin due to a lower rate of ICH, but the rate of NOACs use in many Asian AF is much lower than non-Asian countries due to economic concerns. The purpose of the COhort of antithrOmbotic use and cLinical outcomes in patients with Atrial Fibrillation (COOL-AF) Phase 2 registry is to determine the changes in antithrombotic patterns and the impact on clinical outcomes.

The COOL-AF Phase 2 study is a prospective observational multicenter study of patients with known or newly diagnosed non-valvular AF in Thailand. The aim is a sample size is 3680 patients from 33 centers within a 2-years enrollment timeline. Patients will be follow-up every 6 months until 3 years. The study outcomes were death, ischemic stroke/systemic embolism, major bleeding, myocardial infarction, heart failure, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years and older with atrial fibrillation diagnosed based on a 12-lead ECG or ECG tracing from ambulatory ECG monitoring.

Exclusion Criteria:

1. Patients who have experienced an ischemic stroke within the past 3 months before enrollment.
2. Patients with a platelet count less than 100,000/mm3 or who have myeloproliferative disorders (essential thrombocythemia, chronic myeloid leukemia, polycythemia vera, agnogenic myeloid metaplasia), hyperviscosity syndrome, chronic disseminated intravascular coagulation (DIC), or antiphospholipid syndrome.
3. Patients with a mechanical prosthetic heart valve.
4. Patients with rheumatic mitral stenosis.
5. Patients participating in research projects with concealed treatments.
6. Patients expected to have a life expectancy of less than 3 years due to other diseases, such as cancer or AIDS, as determined from medical records.
7. Pregnancy.
8. Patients unable to follow the treatment plan.
9. Patients who do not consent to participate in the study.
10. Patients who are hospitalized or discharged from the hospital within the past 1 month.Contact/Locations

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-06-02 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of warfarin and NOACs use | 3 years
Rate of ischemic stroke/TIA | 3 years
Rate of systemic embolism | 3 years
Rate of intracranial hemorrhage | 3 years
Rate of major bleeding | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rungroj Krittayaphong, MD,FESC,FACC, Principal Investigator — Division of Cardiology, Department of Medicine, Siriraj Hospital, Mahidol university
Locations (33):
- Thailand (33):
  - Faculty of Meddcine Siriraj Hospital, Mahidol University, Bangkok, Bangkok
  - Faculty of Medicine, Chulalongkorn University,, Bangkok, Bangkok
  - Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Bangkok
  - Faculty of Medicine, Vajira Hospital, Navamindradhiraj University, Bangkok, Bangkok
  - Phramongkutklao College of Medicine, Bangkok, Bangkok
  - Police General Hospital, Bangkok, Bangkok
  - Central Chest Institute of Thailand, Nonthaburi, Changwat Nonthaburi
  - Faculty of Medicine, Prince of Songkla University, Songkhla, Changwat Songkhla
  - Faculty of Medicine, Chiang Mai University,, Chiang Mai, Chiang Mai
  - Bhumibol Adulyadej Hospital, Bangkok
  - Charoen Krung Pracha Rak Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Prapokklao Hospital (Chanthaburi),, Chanthaburi
  - Nakornping Hospital, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Chonburi Hospital, Chon Buri
  - Queen Savang Vadhana Memorial Hospital, Chon Buri
  - Faculty of Medicine, Khon Kaen University, Khon Kaen
  - Lampang Hospital, Lampang
  - Faculty of Medicine, HRH Princess Maha Chakri Sirindhorn Medical Center (MSMC) Srinakharinwirot University, Nakhon Nayok
  - Golden Jubilee Medical Center, Nakhon Pathom
  - Maharat Nakorn Ratchasima Hospital, Nakhon Ratchasima
  - Sawanpracharak Hospital, Nakhon Sawan
  - Faculty of Medicine, Thammasat University, Rangsit Campus, Pathum Thani
  - Buddhachinaraj Hospital, Phitsanulok
  - Faculty of Medicine, Naresuan University, Phitsanulok
  - Vachira Phuket Hospital, Phuket
  - Ratchaburi Hospital, Ratchaburi
  - Sakonnakhon Hospital, Sakon Nakhon
  - Suratthani Hospital, Surat Thani
  - Surin Hospital, Surin
  - Sunpasitthiprasong Hospital, Ubon Ratchathani
  - Udonthani Hospital, Udon Thani

REFERENCES:
- [Derived] Krittayaphong R, Winijkul A, Rungpradubvong V, Apiyasawat S, Phrommintikul A, Chantrarat T, Methavigul K, Chichareon P, Makarawate P, Wongtheptien W, Kaolawanich Y, Lip GYH. The COOL-AF Phase 2 Registry: COhort of Antithrombotic Use and Clinical Outcomes in Atrial Fibrillation Patients. JACC Asia. 2025 Jan 21;5(1):191-202. doi: 10.1016/j.jacasi.2024.10.027. eCollection 2025 Jan. PMID 39896253